CLINICAL TRIAL: NCT02972463
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Dose Ranging Study on the Influence of IgY Max on Inflammatory Markers and the Gut Microbiome
Brief Title: The Influence of IgY Max on Inflammatory Markers and the Gut Microbiome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Igy Nutrition, LLC (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IGYNRPD-150001-RPD01
Record Dates: First submitted 2016-11-18; First posted 2016-11-23 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: Gastrointestinal; Microbiome; Inflammation
MeSH Terms: conditions — Inflammation | interventions — IgY; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): 9 maltodextrin capsules, once daily for 12 weeks
  Interventions: Other: Placebo
- IgY Max Low-Dose (1g IgY Max) (Experimental): 2 Immunoglobulin Y capsules and 7 maltodextrin capsules, once daily for 12 weeks
  Interventions: Dietary Supplement: Immunoglobulin Y
- IgY Max Mid-Dose (2g IgY Max) (Experimental): 4 Immunoglobulin Y capsules and 5 maltodextrin capsules, once daily for 12 weeks
  Interventions: Dietary Supplement: Immunoglobulin Y
- IgY Max High-Dose (4.5g IgY Max) (Experimental): 9 Immunoglobulin Y capsules, once daily for 12 weeks
  Interventions: Dietary Supplement: Immunoglobulin Y

INTERVENTIONS:
Dietary Supplement: Immunoglobulin Y
  Other Names: IgY Max
  Arms: IgY Max High-Dose (4.5g IgY Max); IgY Max Low-Dose (1g IgY Max); IgY Max Mid-Dose (2g IgY Max)
Other: Placebo
  Other Names: Maltodextrin
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the optimal dose of IgY as assessed by changes in the inflammatory marker, C-reactive protein and investigate the effect of IgY on the gut microbiome as assessed by 16s RNA sequencing of fecal samples.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged 18 - 60 (inclusive)
* Self-reported complaints of minor gastrointestinal symptoms (i.e. occasional gas, bloating, etc.)
* Non-smoker, or ex-smoker ≥6 months
* Body mass index 25.0- 34.9kg/m2 (inclusive)
* Female subjects of childbearing potential [i.e. not surgically sterilized or post-menopausal (greater than one year since last menses)] must have negative urine pregnancy test and must be using an effective birth control method
* Willing to avoid alcohol consumption for 24 h prior to every clinic visit
* Willing to maintain their regimens of medications and supplements known to alter GI function (including, but not limited to, iron supplements, calcium, and anti-depressants)
* Willing to maintain a stable body weight, activity level and dietary pattern except for use of the study products, as directed
* Willing and able to provide informed written consent

Exclusion Criteria:

* Pregnancy or lactation, or subject unwilling to take appropriate contraceptives for the duration of the study
* Use of prescription non-steroidal anti-inflammatory drugs (or daily use of over the counter non-steroidal anti-inflammatory drugs >1month), steroids, corticosteroids, or any other prescription anti-inflammatory drugs within 3 months prior to visit 1
* Unstable use (i.e. initiation or change in dose) of antihypertensive medications or thyroid hormone replacement medications within 3 months prior to visit 1
* Use of any weight-loss programs or weight-loss medications (prescription or over-the counter) including, but not limited to, lipase inhibitors, within 3 months prior to visit
* Use of over the counter or prescription laxatives or stool softeners within 1 month prior to baseline (V2)
* Use of antibiotics (other than topical) within 2 months prior to baseline (V2)
* Use of prebiotic supplements (e.g. fructans and galacto-oligosaccharides (FOS, GOS), psyllium, fiber, inulin) or probiotic supplements (i.e. live microorganisms) within 4 weeks of baseline (V2) and consumption of foods fortified with prebiotics (e.g. inulin) or probiotics within 2 weeks of baseline (V2)
* History of blood clotting disorders or use of coagulation-inhibiting drugs (e.g. warfarin)
* Individuals with achlorhydria
* Presence of major diseases such as diabetes, gastrointestinal disease, cardiovascular disease, pancreatic, renal, or liver disease
* Chronic diarrhea or constipation, irritable bowel syndrome, or inflammatory bowel disease
* Abdominal or gastrointestinal surgery within the previous 12 months or planned abdominal or gastrointestinal surgery in the next 4 months
* Recent gastrointestinal food-borne illness (within 1 month prior to visit 1)
* History of neurological disease (e.g. Parkinson's disease, stroke, traumatic brain injury, etc.)
* History of cancer (excluding non-melanoma skin cancer and basal cell carcinoma) in the past 5 years
* Uncontrolled hypertension defined as a seated resting systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg
* Abnormal laboratory test results of clinical significance, including, but not limited to ALT or AST ≥1.5X the upper limit of normal at screening (visit 1)
* Presence or history (past 6 months) of alcohol or drug abuse; alcohol use of >2 standard alcoholic drinks per day
* Extreme dietary habits (e.g. vegan or very low carbohydrate diets)
* Subject has a known allergy or intolerance to the test products or placebo
* Subject is unwilling or unable to abide by the requirements of the protocol
* Any condition that would interfere with the subject's ability to comply with study instructions, might confound the interpretation of the study, or put the subject at risk
* Subject has taken an investigational health product or has participated in a research study within 30 days prior to first study visit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
C-reactive protein | 12 weeks

SECONDARY OUTCOMES:
C-reactive protein | 2 weeks and 4 weeks
Gastrointestinal Symptoms | 2, 4, 8 and 12 weeks
  Total Gastrointestinal Quality of Life Index (GIQLI) score

OTHER OUTCOMES:
Intestinal microbiome | 12 weeks
  As measured by microbial abundance by 16S RNA sequencing of feces
Stool frequency | 12 weeks
  Self-reported number of movements daily averaged over each week
Stool consistency | 12 weeks
  Bristol Stool Scale, self-reported per bowel movement and averaging over each week
Adverse events | 12 weeks
  Number of subjects with a treatment emergent adverse effect

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrasource, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No